CLINICAL TRIAL: NCT07110974
Title: Assessment of Diabetes Distress and Quality of Life in Sohag University Students With Type 1 Diabetes Mellitus
Brief Title: Diabetes Distress and Quality of Life in University Students With Type 1 DM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Dina Abdelnaby Ahmed, assistant lecturer in Family Medicine Luxor University, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Soh-Med-25-7--3MD
Record Dates: First submitted 2025-07-25; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Type 1; Diabetes Distress
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sohag University students with type 1 diabetes mellitus (Other)
  Interventions: Behavioral: Diabetes Distress scale 17 and Quality Of Life Instrument

INTERVENTIONS:
Behavioral: Diabetes Distress scale 17 and Quality Of Life Instrument — questionnaire that assesses the distress resulting from being diabetic patient type 1 and another questionnaire that assesses the quality of life among type 1 diabetic Sohag University students

SUMMARY:
This study aims to encourage and support Sohag University Students with type 1 Diabetes Mellitus (T1DM). It will discover students with poor glycemic control, diabetic retinopathy, and renal complications. In addition to focus on those students suffering from Diabetes Distress (DD) and poor Quality of Life (QOL) due to type 1 Diabetes Mellitus (T1DM).

DETAILED DESCRIPTION:
Data will be collected through personal interviews with type 1 Diabetes Mellitus (T1DM) students using standardized questionnaire. The questionnaire is divided into three sections:

* The first section will gather primarily identification of data such as name, age, gender, father and mother education, order of the student in his/her family, faculty, grade, learning performance, residence; urban or rural, family home or hostile, living alone or with whom, marital status, working, smoking, exercising, history of viral infection as mumps before Diabetes Mellitus (DM), when was first diagnosed with type 1 Diabetes Mellitus (T1DM) and the presentation of the diagnosis, drugs administered for treatment of Diabetes Mellitus (DM) , presence of chronic diseases other than diabetes, history of hospitalization and cause, presence of diabetic complications, and family history of diabetes, we construct the first section according to circumstances in upper Egypt.
* The second section of the questionnaire will be for the assessment of Diabetes Distress (DD) using the valid DDS17 (Diabetes Distress Scale 17) and aims to evaluate distress across four domains: Emotional burden, Physician- related distress, Regimen-related distress, and Interpersonal distress.
* The third section of the questionnaire will be for the assessment of Quality of Life (QOL) using a pre-designed questionnaire called the "Diabetes Quality of Life Instrument" (DQOLI).

ELIGIBILITY:
Inclusion Criteria:

1. Already diagnosed Type 1 diabetes mellitus
2. receiving insulin

Exclusion Criteria:

1. refuses to participate in the study.
2. deaf or mute.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Diabetes Distress Scale 17 (DDS17). Diabetes Quality of Life Instrument | 3 months
  1. Diabetes Distress Scale 17, the degree to which each item may be bothering NOT if the item is true.If that item is not a problem ,circle 1. If it is very bothersome ,circle 6.To score sum the patient's responses and divide by the number of items.
  2. Diabetes Quality of Life Instrument Domain No. of items Range of score for each item Range of score Converted to percentage Domain No of items Range of score Range of score Converted to % Satisfaction (S) 6 for each item 6-30 (S)/30 x 100 Impact (I) 4 4-20 (I)/20 x 100 Worry (W) 3 1-5 3-15 (W)/15 x 100 Total 13 13-65 Total / 65 x 100

IPD SHARING:
Plan to Share IPD: Yes